CLINICAL TRIAL: NCT02892890
Title: Exploratory Study of Predictive Markers of the Therapeutic Response in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy Treated With Intravenous Immunoglobulin
Acronym: EXPRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-24; RCAPHM15_0418 (Registry Identifier: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

ARMS (1):
- patients with CIDP (Experimental)
  Interventions: Procedure: Muscle Magnetic Resonance Imaging (RMI) evaluation; Device: MRI

INTERVENTIONS:
Procedure: Muscle Magnetic Resonance Imaging (RMI) evaluation
Device: MRI

SUMMARY:
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) is an acquired neuropathy characterized by an inflammatory multifocal segmental demyelination. Due to the clinical heterogeneity of this condition and the lack of specific marker that can reliably identify all patients, the diagnosis of CIDP remains difficult. Similarly, there are no clear factors predicting the evolution or the prognosis of the disease. Current treatments are the intravenous immunoglobulin (IVIg), corticoids and plasma exchange; IVIg therapy being the most commonly used. Responses of the patients to the treatments are variable. Thus, it is necessary to identify predictive markers of the therapeutic response of CIDP patients treated by IVIg.

Several potential biomarkers have been proposed recently, but none of them has yet been validated as a predictive criterion for therapeutic response. It is therefore necessary to continue to investigate several biological parameters to identify a reliable biological marker.

In electromyography, the Motor Unit Number Index (MUNIX) technique allows measuring the axonal loss by a precise count of functional motor units. This method, more sensitive than the measure of the Compound Muscle Action Potential (CMAP), is rarely used in CIDP. MUNIX might be a good tool to better characterize the patients and to follow the course of CIDP. It also might be a new sensitive and reliable marker predictive of the therapeutic response.

Magnetic resonance Imaging (MRI) is increasingly used for the assessment of neuromuscular diseases. A recent study on CIDP patients reported a significant decrease of the muscle Magnetisation Transfer Ratio (MTR) compared to healthy subjects, correlated to clinical parameters. The use of advances MRI techniques could allow characterizing the structure and composition of muscle and nerve tissues of CIDP patients. It could also be a mean for identifying potential new markers, largely unexplored until now, that might be sensitive to disease course and/or IVIg response.

The objective of this study is to identify predictive markers of the treatment response of CIDP patients receiving IVIg.

This is a prospective observational exploratory study of a cohort of 30 CIDP patients treated with IVIg and followed-up during one year.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from CIDP
* Fulfilling the EFNS/PNS (European Federation of Neurological Societies / Peripheral nerve Society) 2010 revised criteria
* Treated with IVIg or needed to be treated with IVIg

Exclusion Criteria:

* Patients with a known hypersensitivity to the normal human Ig or one of the constituents of the preparation
* Patients with a known IgA deficiency or with anti-IgA circulating antibodies
* Patients with a change in their immunosuppressive or immunomodulatory treatment in the last 6 months
* Patients with a contraindication for MRI explorations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
decrease of at least one point in the ONLS (Overall Neuropathy Limited Scale) sumscore | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Direction Recherche Clinique APHM
Locations (1):
- APHM, Marseille, France